CLINICAL TRIAL: NCT03448562
Title: Circumferential Pulmonary Vein Isolation Alone Versus. Circumferential Pulmonary Vein Isolation Plus Electrophysiological Substrate Ablation in the Left Atrium During Sinus Rhythm for the Treatment of Non-paroxysmal Atrial Fibrillation
Brief Title: CPVI Alone Versus. CPVI Plus Electrophysiological Substrate Ablation in the LA During SR for the Treatment of Non-PAF
Acronym: STABLE-SR_II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Fudan University (Other); First Affiliated Hospital of Wannan Medical College (Other); The Second Hospital of Hebei Medical University (Other); General Hospital of Shenyang Military Region (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other); Zhongda Hospital (Other); University of Pennsylvania (Other); Southlake Regional Health Centre (Other); German Heart Institute (Other); Asklepios Kliniken Hamburg GmbH (Other); National University Hospital, Singapore (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); National Heart Centre Singapore (Other); Semmelweis University Heart and Vascular Center (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Minglong Chen, Deputy Director of the Department of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-SR-322
Record Dates: First submitted 2017-12-27; First posted 2018-02-28 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Pulmonary Vein Isolation; Catheter Ablation; Substrate Modification
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): CPVI plus electrophysiologic substrate ablation in the left atrium during sinus rhythm (STABLE-SR)
  Interventions: Procedure: CPVI; Procedure: STABLE-SR
- Control Group (Active Comparator): CPVI alone
  Interventions: Procedure: CPVI

INTERVENTIONS:
Procedure: CPVI — ablate around the pulmonary vein orifice
Procedure: STABLE-SR — homogenization of the low voltage zones and elimination of the complex electrograms from the transitional zones during sinus rhythm
  Arms: Study Group

SUMMARY:
The primary objective of this investigation is to compare the efficacy of two different AF ablation strategies in patients with non-paroxysmal AF: CPVI plus electrophysiologic substrate ablation in the left atrium during sinus rhythm (STABLE-SR) and CPVI alone.

DETAILED DESCRIPTION:
BACKGROUND: Atrial fibrillation (AF) is the most common cardiac rhythm disorder, which affects patients' morbidity and mortality. AF ablation has emerged as a promising treatment strategy, offering the possibility of a durable treatment. Currently, there is no general agreement regarding NPAF ablation strategy. Obviously, pulmonary vein isolation is the corner stone for all types of AF ablation. The consensus is that CPVI alone is insufficient for NPAF ablation. However, the recent clinical trials did not show the additional benefits of other substrate modification strategies. Furthermore, the widely used cryo-ablation dilutes the concept that NPAF needs additional substrate modification to further improve the clinical outcome. It seems that CPVI only as the optimal strategy is more commonly accepted for NPAF patients in most of the centers. Based on the results from our pilot study and STABLE-SR trial, we believe that fibrotic substrate modification beyond CPVI is very promising for NPAF ablation, but its superiority over CPVI alone needs a large scaled randomized trial to prove.

AIM OF THE STUDY: The primary objective of this investigation is to compare the efficacy of two different AF ablation strategies in patients with non-paroxysmal AF: CPVI plus electrophysiologic substrate ablation in the left atrium during sinus rhythm (STABLE-SR) and CPVI alone. The primary endpoint is freedom from AF and/or ATs with or without antiarrhythmic drugs (AADs) at 12months after a single-ablation procedure. AF and/or AT occurring in the first 3 months after the ablation (blanking period) was censored. Each episode lasts > 30 seconds. The secondary endpoint are incidence of peri-procedural complications, including stroke, PV stenosis, cardiac perforation, esophageal injury and death; procedure time; fluoroscopy time (including the total fluoroscopy time, during CPVI and after CPVI); the occurrence of the conversion from AF to AT, and its relationship with long-term outcome; the relationship between acute termination of AF and long term outcome.

STUDY DESIGN: This is a randomized, prospective, parallel, single-blind multicenter design. The enrollment target for this investigation is 300 patients. Patients are randomized in a 1:1 fashion into one of the investigation arms: CPVI plus electrophysiologic substrate ablation in the left atrium during sinus rhythm (STABLE-SR) and CPVI alone. Follow-up for these patients includes visits at 3 m, 6 m, 9 m, 12 m.

ELIGIBILITY:
Inclusion Criteria:

* Patients age is 18-80 years;
* Patients with non-paroxysmal AF; non-paroxysmal AF will be defined as a sustained episode lasting > 7 days;
* Patients can sign the written informed consent for the study;
* Patients can endure the required follow-up.

Exclusion Criteria:

* Patients with previous radiofrequency ablation;
* Patients with PLT count less than 80×109/L, or with contraindications to systemic anticoagulation with heparin or Coumadin or a direct thrombin inhibitor;
* Patients with left atrial size ≥ 55 mm (2D echocardiography, parasternal long-axis view);
* Patients with thromboemboli in LA (TEE or MSCT);
* Patients with severe structural cardiac disease (medium or severe mitral regurgitation, DCM, HCM, or other severe valvular heart diseases);
* Patients with abnormal thyroid function;
* Patients with severe liver or renal dysfunction (AST or ALT > 3-fold of upper limit value; the SCr > 3.5 mg/dl or Ccr < 30 ml/min);
* Previous surgery history in last 3 months;
* Patients with life expectancy < 12 months; and
* Patients who are pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from AF and/or ATs with or without antiarrhythmic drugs (AADs) | at least 12 months follow up
  Freedom from AF and/or ATs with or without antiarrhythmic drugs (AADs) at 12months after a single-ablation procedure. AF and/or AT occurring in the first 3 months after the ablation (blanking period) was censored. Each episode lasts > 30 seconds.

SECONDARY OUTCOMES:
Incidence of peri-procedural complications | 1 week after patient enrollment
  stroke, PV stenosis, cardiac perforation, esophageal injury and death
Procedure time | 1 week after patient enrollment
  time that the patient spend in the procedure room
Fluoroscopy time | 1 week after patient enrollment
  the total fluoroscopy time, during CPVI and after CPVI
Occurrence of the conversion from AF to AT | at least 12 months follow up
  the occurrence of the conversion from AF to AT, and its relationship with long-term outcome
Relationship between acute termination of AF and long term outcome | at least 12 months follow up
  the relationship between acute termination of AF and long term outcome

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhang H, Chen N, Bian Q, Yuan M, Yang G, Shen Y, Chen H, Ju W, Li M, Gu K, Wu N, Liu H, Chen M. Persistent atrial fibrillation with left atrial low-voltage area: who benefit from additional modification? Europace. 2025 May 7;27(5):euaf095. doi: 10.1093/europace/euaf095. PMID 40327545
- [Derived] Yang G, Zheng L, Jiang C, Fan J, Liu X, Zhan X, Li J, Wang L, Yang H, Zhu W, Du H, Ma G, Ma W, Kojodjojo P, Chen M; STABLE-SR-II Investigators. Circumferential Pulmonary Vein Isolation Plus Low-Voltage Area Modification in Persistent Atrial Fibrillation: The STABLE-SR-II Trial. JACC Clin Electrophysiol. 2022 Jul;8(7):882-891. doi: 10.1016/j.jacep.2022.03.012. Epub 2022 Apr 27. PMID 35863814